CLINICAL TRIAL: NCT01438073
Title: Elucidating Kisspeptin Physiology by Blocking Kisspeptin Signaling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-P-001564; NCT01862094 (obsolete NCT alias)
Record Dates: First submitted 2011-08-24; First posted 2011-09-21 (Estimated); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Hypogonadotropic Hypogonadism; Healthy Postmenopausal Women; Agonadism
MeSH Terms: conditions — Hypogonadism; Gonadal Dysgenesis | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- kisspeptin, GnRH (Experimental): 24-hour continuous intravenous infusion of kisspeptin 112-121 (12.5-40 mcg/kg/h), single intravenous dose of kisspeptin 112-121 (0.313-13.19 mcg/kg), and single bolus of GnRH (gonadotropin-releasing hormone) (2.5-250 ng/kg)
  Interventions: Drug: kisspeptin 112-121; Drug: GnRH

INTERVENTIONS:
Drug: kisspeptin 112-121 — 24-h continuous intravenous infusion of kisspeptin 112-121 (12.5-40 mcg/kg/h), single intravenous dose of kisspeptin 112-121 (0.313-13.19 mcg/kg)
  Other Names: metastin 45-54
Drug: GnRH — Single intravenous dose of GnRH (2.5-250 ng/kg)
  Other Names: gonadotropin-releasing hormone

SUMMARY:
The investigators are looking for subjects to complete a study on the role of kisspeptin in the reproductive system. Kisspeptin is a naturally occurring hormone in humans that tells the body to produce other reproductive hormones. However, giving someone a continued amount of kisspeptin over a period of time can have the opposite effect and tell the body to, for a short time, stop making hormones needed for reproduction. By giving 24-hour infusions of kisspeptin, the investigators hope to learn more about the role kisspeptin has in the way bodies function normally and the role it has in conditions that affect the reproductive system.

DETAILED DESCRIPTION:
Please contact study staff for a detailed description.

ELIGIBILITY:
A. Healthy Subjects

All healthy subjects will meet the following criteria:

* normal puberty with respect to onset and pace,
* no difficulty with blood draws,
* no prescription medications for at least 2 months with the exception of asthma medication (albuterol only), hypercholesterolemia medication and psychiatric medication,
* no illicit drug use or excessive alcohol consumption (>10 drinks/week),
* no history of a medication reaction requiring emergency medical care,
* normal physical exam and laboratory studies within protocol reference ranges.

Additional criteria based on subject population:

1. Healthy Men:

   * between 21 and 40 years old,
   * normal erectile and ejaculatory function, no history of reproductive disorders,
   * testicular volume >15 ml.
2. Healthy women:

   * between 21 and 40 years old,
   * not breastfeeding or pregnant,
   * menstrual cycles between 25 and 35 days in duration with no more than 5 days variability in cycle duration,
   * no evidence for androgen excess (hirsutism or acne),
3. Healthy postmenopausal women:

   * between 48 and 60 years old,
   * no menstrual periods within the last year,
   * previous history of menstrual cycles between 25 and 35 days in duration, with no more than 5 days variability in cycle duration,
   * if applicable, able to undergo washout from hormone therapy,
   * no evidence for androgen excess (hirsutism or acne),
   * negative screening for Factor V Leiden for those who might receive estradiol treatment as a part of this study.

B. Subjects with Reproductive Disorders

All subjects with reproductive disorders will meet the following criteria:

* all medical conditions stable and well controlled, medications allowed include asthma medication (albuterol only), hypercholesterolemia medication and psychiatric medication,
* no medications known to affect reproductive endocrine function for at least 2 months except for medications used to treat the subject's reproductive condition,
* no history of a medication reaction requiring emergency medical care,
* no illicit drug use or excessive alcohol consumption (>10 drinks/week),
* for women, not breastfeeding or pregnant,
* if applicable, able to undergo appropriate washout from hormone therapy,
* normal physical exam and laboratory studies within protocol reference ranges,

Additional criteria based on subject population:

1. Men and women with hypogonadotropic hypogonadism,

   * 18 years or older,
   * Confirmed diagnosis by low sex steroids in the setting of low or inappropriately normal gonadotropins,
   * If needed, additional labs and imaging tests may be performed.
2. Agonadal men,

   * Between 18 and 60 years old.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Average difference in Luteinizing Hormone (LH) concentration at the beginning and end of kisspeptin infusion | 24 hours

SECONDARY OUTCOMES:
Average difference in testosterone concentration at the beginning and end of kisspeptin infusion (males) | 24 hours
Average difference in estradiol concentration at the beginning and end of kisspeptin infusion (females) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lippincott MF, Chan YM, Rivera Morales D, Seminara SB. Continuous Kisspeptin Administration in Postmenopausal Women: Impact of Estradiol on Luteinizing Hormone Secretion. J Clin Endocrinol Metab. 2017 Jun 1;102(6):2091-2099. doi: 10.1210/jc.2016-3952. PMID 28368443